CLINICAL TRIAL: NCT04776824
Title: Swiss Cardiac Amyloidosis REgistry (Swiss-CARE)
Acronym: B-CARE
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00135
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Amyloid Cardiomyopathy
Keywords: Cardiac Amyloidosis; Tafamidis; CMR feature tracking; Strain; T1 and T2 Mapping; Outcomes
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Genetic testing is a part of the routine diagnostic work-up of TTR amyloidosis patients. Current knowledge suggests that therapy response and clinical outcome may differ in TTR patients suffering from wt-TTR and h-/m-TTR-amyloidosis, respectively. Therefore, the genetic background should also be assessed as part of the registry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed amyloidosis: Confirmed diagnosis of amyloidosis w/wo cardiac involvement

SUMMARY:
Cardiac transthyretin amyloidosis (ATTR), caused by ventricular depositions of misfolded transthyretin, results in an infiltrative cardiomyopathy, progressing from pronounced myocardial wall thickening, diastolic and systolic dysfunction to the development of terminal heart failure. Recently, treatment options for TTR amyloidosis have become available. However costs for therapy are enormous and previous trials were not able to differentiate between patients that might benefit from treatment and those without a need for treatment.

the investigators study aims to determine markers, as assessed by cardiac magnet resonance imaging (CMR) feature tracking (FT) and T1- and T2- mapping, that might reliably indicate disease severity and could help to identify patients that might benefit from (ongoing) TTR stabilization treatment.

DETAILED DESCRIPTION:
Cardiac transthyretin amyloidosis (ATTR), the most common amyloidosis form with cardiac involvement, is caused by tissue deposition of misfolded TTR, a transport Protein for thyroxine and retinol. Ventricular depositions of amyloid fibrils results in an infiltrative cardiomyopathy, progressing from pronounced myocardial wall thickening, to diastolic and systolic dysfunction and finally chronic heart failure.

While treatment options are now available, it remains unclear how to monitor therapy response and disease progression. No makers have been identified that predict outcome prior to initiation of therapy, thus patient selection for therapy remains challenging.

The investigators study will address these issues and will provide systematically assessed CMR data before and over the course of 18 months after therapy initiation. Clinical and laboratory follow-up will be performed every 3-6 months. The investigators study is based on an open, uncontrolled, structured collection of retrospective and prospective data from all patients diagnosed with amyloidosis at the Inselspital Bern with the aim to follow patients undergoing therapy.

The investigators hypothesize that CMR feature tracking (FT) and measures of T1- and T2- mapping, such as extracellular volume (ECV) may better correlate with disease severity and help to identify patients likely to benefit from (ongoing) TTR stabilizing therapy. Beside standard CMR assessments, the investigators will use CMR feature tracking to quantify global and regional myocardial function. FT has proven to be an excellent predictor in various cardiomyopathies.

The proposed study will evaluate the potential of CMR to identify patients likely to benefit from therapy, monitor treatment response and balance individual patient benefit and health care cost.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of amyloidosis w/wo cardiac involvement
* General Consent

Exclusion Criteria:

* Inability to give consent or existence of a written or documented oral refusal of the data subject.<18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of amyloidosis w/wo cardiac involvement
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2001-02-22 (Actual); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
LV (left ventricle) and RV (right ventricle) function as assessed by CMR feature tracking as predictor for MACE (major adverse cardiac event) | 5 years
  Global and regional longitudinal (%), circumferential (%) and radial (%) strain measurements are used to quantify LV and RV function before and after therapy initiation. MACE is defined as a composite of sustained ventricular tachycardia, hospitalization for heart failure and all-cause death.
LV and RV tissue characterization as assessed by T1 and T2 mapping as predictor for MACE | 5 years
  Global and regional tissue characteristics are assessed by repetitive T1 and T2 mapping (global and regional T1 and T2 time (ms)) before and during therapy. MACE is defined as a composite of major cardiovascular endpoints listed above.
Late gadolinium enhancement as predictor for MACE | 5 years
  Global and regional myocardial tissue is characterized by gadolinium contrast agent application. The presence and extent (% and total mass (g)) of late gadolinium enhancement is evaluated as a predictor for MACE.
Extracellular volume (ECV) as predictor for MACE | 5 years
  ECV (%) as a marker of myocardial tissue remodelling is calculated from native and post-contrast T1 mapping and haematocrit before and during therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gräni, MD, PhD, Principal Investigator — Department of Cardiology, University Hospital Bern, Inselspital, Bern
Locations (7):
- Switzerland (7):
  - USB, Basel
  - Department of Cardiology, University Hospital Bern, Inselspital, Bern, Bern
  - HUG, Geneva
  - CHUV, Lausanne
  - LUKS, Lucerne
  - KSSG, Sankt Gallen
  - Stadtspital Triemli, Zurich

IPD SHARING:
Plan to Share IPD: No